CLINICAL TRIAL: NCT04812561
Title: A 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Bronch™ on Respiratory Health
Brief Title: Effects of Bronch™ on Respiratory Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NS_Bronch_01
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Health
Keywords: Respiratory Health; Korean mint; licorice

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronch™ group (Experimental): 2 times a day, 1 pill for 1 time, after breakfast/dinner meal(1,600 mg/day, 800 mg/day as Bronch™)
  Interventions: Dietary Supplement: Bronch™
- Placebo group (Placebo Comparator): 2 times a day, 1 pill for 1 time, after breakfast/dinner meal(1,600 mg/day)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Bronch™ — 2 times a day, 1 pill for 1 time, after breakfast/dinner meal, for 12 week
  Arms: Bronch™ group
Dietary Supplement: placebo — 2 times a day, 1 pill for 1 time, after breakfast/dinner meal, for 12 week
  Arms: Placebo group

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Bronch™(mixture of extraction of Korean mint and licorice) on respiratory health.

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. 60 subjects were randomly divided into Bronch™ group and a placebo group. It is to evaluate the changes in the displayed evaluation items when taking one pill twice a day, in comparison with taking a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80 years at screening
* nonsmoker
* After fully hearing and fully understanding this clinical trials, those who agree to voluntarily decide to participate and to comply with the notice

Exclusion Criteria:

* Participants with clinically significant severe cardiovascular, endocrine, immune, respiratory, liver, biliary, renal and urinary tract, neuropsychiatry, musculoskeletal, inflammatory and hematologic and gastrointestinal disorders
* Participants who have Body Mass Index(BMI) less than 18.5 kg/m^2 or more than 35 kg/m^2
* Participants who have taken medication or dietary supplements related to the respiratory disease within 1 months prior to screening
* Participants with a history of antipsychotic medication use within 3 months prior to the screening examination
* Participants who alcoholic or drug abuse suspected
* Participants who have participated in the other human trials within 3 months before the screening test
* Laboratory test by show the following results

  * AST, ALT > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dL
* Pregnancy or breast feeding
* Patients who are judged ineligible to participate in the trial by the principal investigator for other reasons, including laboratory test outcomes

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Changes of CAT{Chronic obstructive pulmonary disease(COPD) Assessment Test} scores | screening, 6, 12 week
  CAT were measured in study screening, visit 2(6 week), visit 3(12 week). CAT was developed for use as a way to assess the quality of life of COPD patients, consisting of eight items, each of which evaluates 0 to 5 points, and the sum of all eight item scores is the CAT score. The best quality of life is 0 points, and the worst is 40 points.
Changes of BCSS(Breathlessness, Cough, and Sputum Scale) scores | 0, 6, 12 week
  BCSS were measured in study visit 1(0 week), visit 2(6 week), visit 3(12 week). BCSS is a scale for evaluating symptoms of Breathlessness, cough, and sputum, which is a major symptom of COPD(Chronic obstructive pulmonary disease), and symptoms of Breathlessness, cough, and sputum are evaluated in five stages.
  <Breathlessness, sputum> 0: never, 1: rare, 2: occasionally, 3: often, 4: almost always <Cough> 0: never, 1: a little hard, 2: moderate extent of hard, 3: over moderate extent of hard, 4: serious hard

SECONDARY OUTCOMES:
FVC(Forced vital capacity) | screening, 12 week
  The Forced vital capacity(FVC) was measured Flow rate discharged during the hard-working unit before and after the intervention.
FEV1(Forced expiratory volume in 1 second) | screening, 12 week
  The Forced expiratory volume in 1 second(FEV1) was assessed before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea